CLINICAL TRIAL: NCT05863143
Title: Effectiveness of Nutritional and Exercise Intervention on Reducing Risk of Falls Among Community Dwelling Older Adults in Selangor
Brief Title: Intervention on Reducing Risk of Falls Among Community Dwelling Older Adults in Selangor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Chan Yoke Mun, Professor, Universiti Putra Malaysia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UPM11062022
Record Dates: First submitted 2022-12-21; First posted 2023-05-17 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Fall
Keywords: risk of falls; nutrition; exercise; TUG; intervention; community dwelling older adults
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Subjects in the intervention group are required to involve in 12 sessions of nutrition education program and prescribed exercise program during the 12 weeks intervention period. Generally, respondents in the intervention group will received the developed educational materials and exercise diary as guide during this period.
  Interventions: Behavioral: Nutritional and Exercise
- Control Group (No Intervention): Subjects required to continue with usual lifestyle (eating habits and exercise pattern) for 12 weeks. Tips on healthy eating and active living, which are suitable for them will be provided.
  When the study is completed (after 12 weeks), they will receive the same intervention activities as the intervention group.

INTERVENTIONS:
Behavioral: Nutritional and Exercise — Provide Nutritional Education Program and Falls Module Exercise (FME) to the intervention group
  Arms: Intervention Group

SUMMARY:
Falls is a major concern in geriatrics due to its high prevalence and various adverse health complications among elderly population. Risk of falls can be reduced by improving nutritional status and increase the level of physical activity. Besides, knowledge regarding risk of falls, nutrition and exercise are important in reducing the risks of falls. Therefore, this study aims to develop, implement and evaluate the effectiveness of a nutritional education and exercise intervention among community dwelling older adults in Selangor.

DETAILED DESCRIPTION:
General Objective: To develop, implement and evaluate the effectiveness of nutrition education and exercise intervention on risk of fall among older person in Selangor.

Specific Objectives:

* To determine the risk of falls among the older adults.
* To determine the dietary intake, anthropometric parameters (body mass index, mid upper arm circumference, calf circumference, body fat percentage and skeletal muscle mass), nutritional status, level of physical activity, functional status, perceived quality of life, risk of sarcopenia, level of knowledge, attitude and practice (KAP) towards falls' risk reduction, nutrition and exercise among the older adults.
* To identify the factors determining risk of falls among older adults.
* To evaluate the implementation process of the nutrition education and exercise intervention program (attendance and feedback of the program).
* To determine the mean differences in risk of falls, dietary intake, anthropometric parameters, nutritional status, physical activity, functional status, perceived quality of life, risk of sarcopenia and knowledge, attitude and practice (KAP) towards falls' risks reduction, nutrition and exercise between intervention and control groups before and after intervention.

The proposed study location is in Selangor. This is a randomized wait-list controlled trial for 3 months (12 weeks) among community dwelling older adults in Selangor. A two-stage sampling design will be applied. Firstly, a random sampling will be applied to select two districts from Selangor. This is followed by a purposive sampling to recruit eligible subjects according to inclusion criteria.

Subjects will be recruited from free living older adults residing in Selangor through various community settings including including affiliations of National Council of Senior Citizens Organisations Malaysia (NACSCOM), University of Third Age (U3A) and Alzheimer's Disease Foundation Malaysia (ADFM).

Subjects will be allocated randomly into 2 groups:

Group 1: Intervention group (nutrition education + exercise intervention) Group 2: Control group (no intervention)

which total of 100 eligible subjects will be recruited, with 50 subjects are needed in respective groups.

This study will use a set of questionnaires to obtain information on personal information, anthropometry data, nutritional status, level of physical activity, functional status, sleep quality, quality of life, risk of falls, risk of sarcopenia and KAP on falls' risk reduction, nutrition and exercise based on appropriate instruments. Assessments will be performed at baseline (week 0), mid-way (week 6) and post-intervention (after week 12).

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 60 years old to 80 years old in Malaysia
* Able to ambulate without personal assistance
* Able to read and write

Exclusion Criteria:

* Self-reported chronic diseases (severely poorly control diabetics and hyperlipidemia, heart-related disease, Chronic obstructive pulmonary disease, osteoarthritis, osteoporosis, stroke, cancer, asthma, renal dysfunction, terminally ill that may limit participations in physical activity)
* Any sustained fracture or undergoing surgery (hip, vertebrata) in past six months
* Bedridden
* Sensory impairment (visual & hearing) that will interfere with communication
* Anyone who participated in similar program before

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-23 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Mean Changes in Risk of Falls | Assessments will be performed at Baseline (Week 0), mid-intervention (Week 6) and Post-Intervention (Week 12)
  Risk of falls of the respondents will be determined using Timed Up and Go (TUG) test, Five Times Sit to Stand Test (5XSST) and 30 Second Sit to Stand Test (30CST). For the Timed Up and Go (TUG) test, respondents will be timed while they rise from an arm- chair, walk at a comfortable and safe pace to a line on the floor three meters away (10 feet), turn and walk back to the chair and sit down again. The respondents will walk through the test once before being timed to become familiar with the test.
Mean Changes in Risk of Falls | Assessments will be performed at Baseline (Week 0), mid-intervention (Week 6) and Post-Intervention (Week 12)
  Besides assessing risk of falls using Timed Up and Go (TUG) test, risk of falls of the respondents will be determined using Five Times Sit to Stand Test (5XSST) and 30 Second Sit to Stand Test (30CST). Five Times Sit to Stand Test is performed to determine time taken for respondent to shift five times from a seated to a standing posture.
Mean Changes in Risk of Falls | Assessments will be performed at Baseline (Week 0), mid-intervention (Week 6) and Post-Intervention (Week 12)
  Besides assessing risk of falls using Timed Up and Go (TUG) test and Five Times Sit to Stand Test, risk of falls of the respondents will be determined using 30 Second Sit to Stand Test (30CST). For 30 Second Sit to Stand Test, respondents are required to sit straight on a chair with arms are crossed at the wrists and held in front of the chest. The respondents are encouraged to complete as many full stands as possible within 30 seconds.

SECONDARY OUTCOMES:
Mean Changes in Skeletal Muscle Mass | Assessments will be performed at Baseline (Week 0), mid-intervention (Week 6) and Post-Intervention (Week 12)
  Risk of sarcopenia among the older adults will be determined according to the Asian Working Group for Sarcopenia (AWGS) Criteria 2014. This is to be ascertained on muscle mass, handgrip strength and gait speed. The skeletal muscle mass will be accessed in gram using the InBody Body Impedance Analyzer (BIA) (S10 model) to help derive the skeletal muscle mass index. Grip strength will be measured using a Jamar dynamometer. Three measurements of hand grip strength will be taken for the dominant hand, with the mean value of three measurements to be recorded. For gait speed, respondents are required to walk on six meters of a straight path (about 20 feet) with time taken will be taken. The faster time of two trials will be recorded.
Mean Changes in Handgrip Strength | Assessments will be performed at Baseline (Week 0), mid-intervention (Week 6) and Post-Intervention (Week 12)
  Risk of sarcopenia among the older adults will be determined according to the Asian Working Group for Sarcopenia (AWGS) Criteria 2014. This is to be ascertained on muscle mass, handgrip strength and gait speed. Grip strength will be measured in kilograms (kg) using a Jamar dynamometer. Three measurements of hand grip strength will be taken for the dominant hand, with the mean value of three measurements to be recorded.
Mean Changes in Gait Speed | Assessments will be performed at Baseline (Week 0), mid-intervention (Week 6) and Post-Intervention (Week 12)
  Risk of sarcopenia among the older adults will be determined according to the Asian Working Group for Sarcopenia (AWGS) Criteria 2014. This is to be ascertained on muscle mass, handgrip strength and gait speed. For gait speed, respondents are required to walk on six meters of a straight path (about 20 feet) with time taken will be taken. The faster time of two trials will be recorded.
Mean Changes in Energy Intake | Assessments will be performed at Baseline (Week 0), mid-intervention (Week 6) and Post-Intervention (Week 12)
  Three-day 24 hours dietary recall will be used to obtain the dietary data of older adults. Respondents are required to recall the food and beverages taken in the previous 24 hours for two weekdays and one weekend day. Time of consumption, type of food, serving size and size of household units will be recorded in the diet recall form through face-to-face interview. Household measures such as plates, bowls and spoons of different sizes will be used during data collection to quantify food intake of the respondents. Nutritionist Pro will be used to analyze energy intake in kcal with the use of several databases including Malaysian Food Composition Database, USDA Standard Reference Database, Food and Nutrient Database for Dietary Studies and others.
Mean Changes in Protein Intake | Assessments will be performed at Baseline (Week 0), mid-intervention (Week 6) and Post-Intervention (Week 12)
  Three-day 24 hours dietary recall will be used to obtain the dietary data of older adults. Respondents are required to recall the food and beverages taken in the previous 24 hours for two weekdays and one weekend day. Time of consumption, type of food, serving size and size of household units will be recorded in the diet recall form through face-to-face interview. Household measures such as plates, bowls and spoons of different sizes will be used during data collection to quantify food intake of the respondents. Nutritionist Pro will be used to analyze protein intake in gram (g) with the use of several databases including Malaysian Food Composition Database, USDA Standard Reference Database, Food and Nutrient Database for Dietary Studies and others.
Mean Changes in Calcium Intake | Assessments will be performed at Baseline (Week 0), mid-intervention (Week 6) and Post-Intervention (Week 12)
  Three-day 24 hours dietary recall will be used to obtain the dietary data of older adults. Respondents are required to recall the food and beverages taken in the previous 24 hours for two weekdays and one weekend day. Time of consumption, type of food, serving size and size of household units will be recorded in the diet recall form through face-to-face interview. Household measures such as plates, bowls and spoons of different sizes will be used during data collection to quantify food intake of the respondents. Nutritionist Pro will be used to analyze calcium intake in gram (g) with the use of several databases including Malaysian Food Composition Database, USDA Standard Reference Database, Food and Nutrient Database for Dietary Studies and others.
Mean Changes in Vitamin D Intake | Assessments will be performed at Baseline (Week 0), mid-intervention (Week 6) and Post-Intervention (Week 12)
  Three-day 24 hours dietary recall will be used to obtain the dietary data of older adults. Respondents are required to recall the food and beverages taken in the previous 24 hours for two weekdays and one weekend day. Time of consumption, type of food, serving size and size of household units will be recorded in the diet recall form through face-to-face interview. Household measures such as plates, bowls and spoons of different sizes will be used during data collection to quantify food intake of the respondents. Nutritionist Pro will be used to analyze vitamin D intake in microgram (mcg) with the use of several databases including Malaysian Food Composition Database, USDA Standard Reference Database, Food and Nutrient Database for Dietary Studies and others.
Mean Changes in Weight | Assessments will be performed at Baseline (Week 0), mid-intervention (Week 6) and Post-Intervention (Week 12)
  Seca 803 Digital Weight Scale will be used to measure body weight of the respondents in light clothing (without shoes) to the nearest 0.1 kilogram, using standardized protocol.
Mean Changes in Height | Assessments will be performed at Baseline (Week 0), mid-intervention (Week 6) and Post-Intervention (Week 12)
  Standing height of the respondents will be taken using SECA portable stadiometer (SECA-213 model) to the nearest 0.1 centimeter with the subject standing barefoot. The head will be kept in the Frankfurt plane and heels checked to make sure they were on the platform. Respondents who are found to have kyphosis problem or difficulty to stand straight will be not taken their standing height but replaced with alternative height (demi-span) measurement.
Mean Changes in calf-circumference | Assessments will be performed at Baseline (Week 0), mid-intervention (Week 6) and Post-Intervention (Week 12)
  Calf circumference will be measured using a flexible non-stretchable tape (SECA-201 model). This is a recognized anthropometric parameter to indicate muscle loss especially in the lower limb and considered a pertinent marker of the nutritional status in the elderly. During measurement, the tape will be wrapped comfortably around the calf (non-dominant leg) at the widest part while respondents are sitting down and recorded to the nearest 0.1cm.
Mean Changes in Physical Activity Level | Assessments will be performed at Baseline (Week 0), mid-intervention (Week 6) and Post-Intervention (Week 12)
  The level of physical activity among the respondents will be assessed using the Rapid Assessment of Physical Activity (RAPA), which is a user friendly and validated tool to assess levels of physical activity among older people aged 50 and above. It is made up of nine "Yes" or "No" questions to evaluate the amount and intensity of physical activity of the respondents. It is divided into two components, namely an assessment of aerobic activity from sedentary to moderate and vigorous sports as well as an evaluation of activities that increase strength and flexibility. For the first component on assessment of aerobic activity, respondents are required to choose one question which reflected their level of physical activity with affirmative response. The scores for aerobic activity would be increased if the amount, frequency and intensity of physical activity increased. The scores for these components ranged from 1 to 7 points.
  Two questions will be developed for the assessment on strength
Mean Changes in Nutritional Status | Assessments will be performed at Baseline (Week 0), mid-intervention (Week 6) and Post-Intervention (Week 12)
  Nutritional status will be assessed using the short form of the Mini Nutritional Assessment (MNA-SF). The MNA-SF is an effective, easily administered tool designed to identify older adults who have or are at risk of developing malnutrition. This short-standardized questionnaire comprises six questions about food decline, weight loss in the last three months, mobility, actual disease/distress, psychological situation, and additionally anthropometric measures (body mass index or calf circumference). MNA-SF scores will be categorized into three different categories where score below eight indicates malnutrition, 8-11 indicates at risk of malnutrition and 12- 14 represents well-nourished status.
Mean Changes in Functional Status | Assessments will be performed at Baseline (Week 0), mid-intervention (Week 6) and Post-Intervention (Week 12)
  The well-established Lawton Instrumental Activities of Daily Living (IADL) questionnaire will be used to assess the respondents' ability to perform eight daily activities (i.e. ability to use telephone, shopping, preparing meals, housekeeping, doing laundry, using public transport, taking medications, and handling finances). Presence of 'functional disability' will be defined as having difficulty or needing help in at least one of these 8 items IADL activities, while normal functioning will be defined if one can perform all 8 activities independently.
Mean Changes in Quality of Life | Assessments will be performed at Baseline (Week 0), mid-intervention (Week 6) and Post-Intervention (Week 12)
  The perceived quality of life of the respondents will be determined using Older Person Quality of Life (OPQOL) Questionnaire. This questionnaire consists of 35 statements with the participant being asked to indicate the extent to which he/she agrees with every single statement by choosing one of five possible options among "strongly disagree", "disagree", "neither agree nor disagree", "agree" and "strongly agree". Each of the five possible answers is given a score of 1 to 5 so that higher scores indicate a better QOL. Thus, the total score ranges from 35 (the worst possible QOL) to 175 (the best possible QOL). The 35 statements of the questionnaire consider the following aspects of QOL: life overall, health (score range 4-20), social relationships and participation, independence, control over life and freedom, home and neighbourhood, psychological and emotional well-being, financial circumstances, leisure, activities and religion.
Mean Changes in Knowledge, Attitude and Practice on Falls' risk reduction, nutrition and exercise Questionnaire | Assessments will be performed at Baseline (Week 0) and Post-Intervention (Week 12)
  Knowledge, attitude and practice on falls, nutrition and exercise of the respondents will be assessed sing a self-developed questionnaire. This questionnaire consists of 9 domains and 101 items related to KAP on Falls reduction, nutrition and exercise and have been undergone content and face validities. Higher score represent better knowledge, attitude and practice.
Mean Changes in Sleep Quality | Assessments will be performed at Baseline (Week 0), mid-intervention (Week 6) and Post-Intervention (Week 12)
  Sleeping quality of the respondents will be determined using Pittsburgh Sleep Quality Index (PSQI). PSQI is a structured, self-administered questionnaire that measures retrospective sleep quality and disturbances within the past month. The 7 self-rated questions assess a wide variety of factor related to sleep quality, including estimates of sleep duration and latency. These 7 items are grouped into five component scores, each weighted equally on a 0-3 scale. The five component scores are then summed to yield a sleep quality index score, which has a range of 0-15, with higher scores indicate worse sleep quality. The five components are subjective sleep quality, sleep latency, sleep duration, sleep disturbances and use of sleep medication.

CONTACTS AND LOCATIONS:
Overall Officials: Yoke Mun Chan, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Universiti Putra Malaysia, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No